CLINICAL TRIAL: NCT00840801
Title: SINGLE-BLIND, RANDOMIZED, PHASE III B STUDY IN CHILDREN AGED 1 - 11 YEARS TO INVESTIGATE THE IMMUNOGENICITY, SAFETY AND INTERCHANGEABILITY OF TWO TICK-BORNE ENCEPHALITIS (TBE) VACCINES ADMINISTERED ACCORDING TO A CONVENTIONAL SCHEDULE
Brief Title: Immunogenicity, Safety and Interchangeability of Two Tbe Vaccines Administered According to a Conventional Schedule in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Single | Purpose: Prevention
Other Study IDs: 700801; B9371022 (Other: Alias Study Number); 2008-002691-10 (EudraCT Number); EUDRACT NUMBER: 2008-002691-10
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Encephalitis, Tick-Borne
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects receive three vaccinations with a paediatric TBE vaccine according to the conventional vaccination schedule.
  Interventions: Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated)
- 2 (Experimental): Subjects receive three vaccinations with a paediatric TBE vaccine according to the conventional vaccination schedule.
  Interventions: Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated)

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated) — Subjects receive three vaccinations with FSME-IMMUN 0.25ml Junior on days 0, 28 and 360
  Arms: 1
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated) — Subjects receive two vaccinations with Encepur 0.25ml Children on days 0 and 28 and a third vaccination with FSME-IMMUN 0.25ml Junior on day 360.
  Arms: 2

SUMMARY:
The objective of this study is to assess the immunogenicity, safety and interchangeability of two different TBE vaccines in children aged 1-11 years, the first and second vaccination with either FSME-IMMUN 0.25ml Junior or Encepur 0.25ml Children and the third vaccination with FSME-IMMUN 0.25 ml Junior only, administered according to the conventional schedule (0, 28 and 360 days).

ELIGIBILITY:
Inclusion Criteria:

Male and female children will be eligible for participation in this study if:

* they are aged >= 1 years (from the 1st birthday) to 11 years (to the last day before the 12th birthday) at screening;
* their parents / legal guardians provide written informed consent;
* children provide written assent to the study according to age and capacity of understanding;
* their parents/guardians understand the nature of the clinical study and will comply with the requirements of the protocol (e.g., completion of the Subject Diary, return for follow-up visits);
* they are generally healthy, (i.e. the physician would have no reservations vaccinating with a TBE vaccine outside the scope of a clinical study);
* provide a negative pregnancy test result at the first medical examination (if the subject is a female and capable of bearing children).

Exclusion Criteria:

Subjects will be excluded from participation if:

* they have a history of any previous TBE vaccination;
* they have a history of TBE infection;
* they have a history of infection with other flaviviruses;
* they have a history of vaccination against yellow fever and/or Japanese B encephalitis;
* they have a history of severe allergic reactions, in particular a known sensitivity or allergy to any components of the vaccines;
* they are suffering from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immunological functions;
* they have received any blood product or immunoglobulins within 90 days prior to study entry;
* they are known to be Human Immunodeficiency Virus (HIV) positive (an HIV test is not required specifically for the purpose of this study);
* they have a functional or surgical asplenia;
* they have a rash or other dermatological condition at the injection site which could interfere with injection site reaction evaluation;
* they were administered an investigational product within six weeks prior to study start or are concurrently participating in another clinical study that includes the administration of an investigational product;
* they are pregnant or breastfeeding (if a female subject);
* they or their parents/legal guardian(s) are in a dependent relationship with the study investigator or with a study team member. Dependent relationship includes close relatives (i.e., children or grandchildren, partner/spouse, siblings) as well as employees of the investigator or site conducting the study.
* Subjects who have an acute illness with or without elevated body temperature (>=37.5°C) within 3 days prior to the scheduled first vaccination will not be vaccinated. Subjects may be included at a repeat visit provided that (1) the illness has resolved (body temperature < 37.5 °C), (2) the repeat visit is no more than 14 calendar days after the Screening Visit, and (3) the center is still open for recruitment.
* If subjects have received antipyretics within 4 hours prior to the scheduled time of vaccination, the vaccination should be performed at a later date, as long as the center is still open for recruitment.
* Subjects who received any live vaccine within 4 weeks or any inactivated vaccine within 2 weeks prior to the scheduled first study vaccination will not be vaccinated until an interval of 4 or 2 weeks, respectively, has passed, provided the center is still open for recruitment.
* If a subject was bitten by a tick within 4 weeks prior to the scheduled first or second vaccination, the vaccination must be postponed until an interval of 4 weeks has passed.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2009-02-06 (Actual); Primary Completion 2010-05-20 (Actual); Study Completion 2010-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Baxter Bioscience Investigator, Principal Investigator — Baxter BioScience
Locations (6):
- Austria (2):
  - Unterer Graben 2, Eferding, Upper Austria
  - Grieskirchnerstr.17, Wels, Upper Austria
- Czechia (4):
  - Private surgery of General Practitioner for children and juveniles, Havlíčkův Brod
  - University Hospital Hradec Kralove, Vaccinal center, Clinic of infectious diseases, Sokolská 581, Hradec Králové
  - Private surgery of General Practitioner for children and juveniles, Pardubice
  - Chemiku 129, Pardubice-Polabiny

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=700801&StudyName=Immunogenicity%2C%20safety%20and%20interchangeability%20of%20two%20tbe%20vaccines%20administered%20according%20to%20a%20conventional%20schedule%20in%20children

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted from 06 February 2009 to 20 May 2010 in Austria and Czech Republic.
Groups:
- Part A: FSME-IMMUN: Participants received FSME-IMMUN (FSME-IMMUN Junior) at Day 0 and 28 as first and second vaccination according to the conventional immunization schedule.
- Part A: Encepur: Participants received Encepur (Encepur Children) at Day 0 and 28 as first and second vaccination according to the conventional immunization schedule.
- Part B: FSME-IMMUN: Participants received FSME-IMMUN (FSME-IMMUN Junior) at Day 360 as third vaccination in period 2.
Period: Part A: Screening- Day 28 Postdose 2
Arm/Group | Part A: FSME-IMMUN | Part A: Encepur | Part B: FSME-IMMUN
Started | 150 | 152 | 0
Completed | 149 | 152 | 0
Not Completed | 1 | 0 | 0
Not completed — Screen failure | 1 | 0 | 0
Period: Part B:Day 28 Postdose2-Day 28 Postdose3
Arm/Group | Part A: FSME-IMMUN | Part A: Encepur | Part B: FSME-IMMUN
Started | 0 (All participants received FSME-IMMUN. Thus, the participant flow for this arm has not been reported.) | 0 (All participants received FSME-IMMUN. Thus, the participant flow for this arm has not been reported.) | 301 (Participants received FSME-IMMUN (encompassing both Part A: FSME-IMMUN and Part A: Encepur arms).)
Completed | 0 (All participants received FSME-IMMUN. Thus, the participant flow for this arm has not been reported.) | 0 (All participants received FSME-IMMUN. Thus, the participant flow for this arm has not been reported.) | 297 (Participants received FSME-IMMUN (encompassing both Part A: FSME-IMMUN and Part A: Encepur arms).)
Not Completed | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1
Not completed — Refused blood draw | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received the third vaccination of FSME-IMMUN, after first 2 doses of FSME-IMMUN or Encepur and had documented adverse event information at least immediately afterwards.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: FSME-IMMUN | Part A: Encepur | Total
Number analyzed (Participants) | 150 | 152 | 302
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days- 23 months) | 50 | 50 | 100
  Children (2-11 years) | 100 | 102 | 202
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 74 | 151
  Male | 73 | 78 | 151

OUTCOME MEASURES:

1. Primary Outcome: Seropositivity Rate as Determined by Neutralization Test (NT) 28 Days After the Second Vaccination
Description: Percentage of participants achieving NT titer greater than or equal to (>=) 10.
Time Frame: 28 days after Vaccination 2
Population: Per-protocol analysis set included eligible participants who received first and second vaccination; had negative baseline values in NT; had immunogenicity measurements available at baseline; 28 days after second vaccination and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- FSME-IMMUN: It Included participants who received FSME-IMMUN during the first and second vaccination.
- Encepur: It Included participants who received Encepur during the first and second vaccination.
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 127 | 134
Percentage of participants | 100 [97.1 to 100] | 97.8 [93.6 to 99.5]
Statistical Analysis 1: Comparison: FSME-IMMUN vs Encepur; Non-inferiority Test on Seropositive Response Rate; Test type: Non-Inferiority or Equivalence — A stratified score test was used to test the non-inferiority with a margin of -10% at 2.5% type I error (one-sided); p < 0.001, Stratified score test

2. Secondary Outcome: Seropositivity Rate Determined by NT 180 Days After the First Vaccination and 28 Days After the Third Vaccination
Description: Percentage of participants with NT titer >=10. Here, "number of participants analyzed" signifies total number of participants included in the modified intent-to-treat (mITT) population and "Number Analyzed" signifies number of participants who were evaluable at specified timeframe.
Time Frame: 180 days after the Vaccination 1, 28 days after the Vaccination 3
Population: mITT analysis set included eligible participants who fulfilled all inclusion and exclusion criteria, received first and second vaccination, had no positive baseline values in ELISA(IMMUNOZYM FSME ELISA and Enzygnost TBE ELISA)and NT, had immunogenicity measurements available at baseline and 28 days after second vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- FSME-IMMUN: It Included participants who received FSME-IMMUN during the first and second vaccination, received FSME-IMMUN at Day 360 as third vaccination.
- Encepur: It Included participants who received Encepur during the first and second vaccination, received FSME-IMMUN at Day 360 as third vaccination.
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 149 | 152
Percentage of participants
  180 Days after Vaccination 1: number analyzed (Participants) | 129 | 133
  180 Days after Vaccination 1 | 95.3 [90.2 to 98.3] | 91 [84.8 to 95.3]
  28 Days after Vaccination 3: number analyzed (Participants) | 128 | 132
  28 Days after Vaccination 3 | 100 [97.2 to 100] | 100 [97.2 to 100]

3. Secondary Outcome: Seropositivity Rate Determined by ELISA 28 Days After the Second Vaccination, 180 Days After the First Vaccination and 28 Days After the Third Vaccination
Description: Percentage of participants with IMMUNOZYM ELISA >126 Vienna Units per milliliter (VIEU/mL) or Enzygnost ELISA >10.32 Units per milliliter (U/mL). Here, "Number Analyzed" signifies number of participants who were evaluable at the specified timeframe.
Time Frame: 28 days after Vaccination 2, 180 days after the Vaccination 1, 28 days after the Vaccination 3
Population: mITT analysis set included eligible participants who fulfilled all inclusion and exclusion criteria, received first and second vaccination, had no positive baseline values in ELISA (IMMUNOZYM FSME ELISA and Enzygnost TBE ELISA) and NT, had immunogenicity measurements available at baseline and 28 days after second vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 149 | 152
percentage of participants
  180 Days after Vaccination 1: number analyzed (Participants) | 142 | 146
  180 Days after Vaccination 1 | 95.1 [90.1 to 98] | 81.5 [74.2 to 87.4]
  28 Days after Vaccination 2: number analyzed (Participants) | 143 | 148
  28 Days after Vaccination 2 | 100 [97.5 to 100] | 97.3 [93.2 to 99.3]
  28 Days after Vaccination 3: number analyzed (Participants) | 141 | 145
  28 Days after Vaccination 3 | 100 [97.4 to 100] | 100 [97.5 to 100]

4. Secondary Outcome: Antibody Response Measured by NT 28 Days After the Second Vaccination, 180 Days After the First Vaccination and 28 Days After the Third Vaccination
Description: Geometric mean of antibody response measured by NT. Here, "Number Analyzed" signifies number of participants who were evaluable at the specified timeframe.
Time Frame: 28 days after Vaccination 2, 180 days after Vaccination 1, 28 days after Vaccination 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 149 | 152
titer
  180 Days after Vaccination 1: number analyzed (Participants) | 129 | 133
  180 Days after Vaccination 1 | 39.7 [34.4 to 45.8] | 25 [21.3 to 29.4]
  28 Days after Vaccination 2: number analyzed (Participants) | 129 | 135
  28 Days after Vaccination 2 | 236.8 [199.6 to 281] | 118.8 [97.5 to 144.9]
  28 Days after Vaccination 3: number analyzed (Participants) | 128 | 132
  28 Days after Vaccination 3 | 538.2 [499.2 to 580.2] | 521.3 [476.6 to 570.2]

5. Secondary Outcome: Antibody Response Measured by ELISA 28 Days After the Second Vaccination, 180 Days After the First Vaccination and 28 Days After the Third Vaccination
Description: Geometric mean of antibody response measured by IMMUNOZYM ELISA (VIEU/mL) and Enzygnost ELISA (U/mL). Here, "Number Analyzed" signifies number of participants who were evaluable at specified timeframe for the specified ELISA assay.
Time Frame: 28 days after Vaccination 2, 180 days after Vaccination 1, 28 days after Vaccination 3
Population: mITT analysis set included eligible participants who fulfilled all inclusion and exclusion criteria, received first and second vaccination, had no positive baseline values in ELISA (IMMUNOZYM FSME ELISA and Enzygnost TBE ELISA) and NT, had immunogenicity measurements available at baseline and 28 days after the second vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 149 | 152
titer
  IMMUNOZYM: 180 Days after Vaccination 1: number analyzed (Participants) | 142 | 147
  IMMUNOZYM: 180 Days after Vaccination 1 | 493.7 [436.5 to 558.5] | 161.2 [140.5 to 184.9]
  IMMUNOZYM: 28 Days after Vaccination 2: number analyzed (Participants) | 143 | 149
  IMMUNOZYM: 28 Days after Vaccination 2 | 3026.3 [2652.2 to 3453.2] | 678 [561.2 to 819.2]
  IMMUNOZYM: 28 Days after Vaccination 3: number analyzed (Participants) | 141 | 146
  IMMUNOZYM: 28 Days after Vaccination 3 | 11292.9 [9693.5 to 13156.3] | 10508.6 [8208.4 to 13453.3]
  Enzygnost: 180 Days after Vaccination 1: number analyzed (Participants) | 148 | 149
  Enzygnost: 180 Days after Vaccination 1 | 47.9 [41.4 to 55.4] | 26.7 [22.5 to 31.6]
  Enzygnost: 28 Days after Vaccination 2: number analyzed (Participants) | 149 | 151
  Enzygnost: 28 Days after Vaccination 2 | 163.3 [152.8 to 174.5] | 93.7 [81.6 to 107.5]
  Enzygnost: 28 Days after Vaccination 3: number analyzed (Participants) | 147 | 148
  Enzygnost: 28 Days after Vaccination 3 | 682.2 [579.6 to 802.9] | 673.2 [533.4 to 849.7]

6. Secondary Outcome: Fold Increase of Antibody Response Measured by NT 28 Days After the Second Vaccination, 180 Days After the First Vaccination and 28 Days After the Third Vaccination as Compared to Baseline
Description: Geometric mean of fold increase of antibody response measured by NT from day 0 to specified timeframe. Here, "Number Analyzed" signifies number of participants who were evaluable at specified timeframe.
Time Frame: 28 days after Vaccination 2, 180 days after Vaccination 1, 28 days after Vaccination 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 149 | 152
fold rise
  180 Days after Vaccination 1: number analyzed (Participants) | 129 | 133
  180 Days after Vaccination 1 | 7.9 [6.8 to 9.1] | 5 [4.2 to 5.8]
  28 Days after Vaccination 2: number analyzed (Participants) | 129 | 135
  28 Days after Vaccination 2 | 46.9 [39.5 to 55.8] | 23.6 [19.4 to 28.8]
  28 Days after Vaccination 3: number analyzed (Participants) | 128 | 132
  28 Days after Vaccination 3 | 106.7 [98.5 to 115.5] | 103.5 [94.6 to 113.2]

7. Secondary Outcome: Fold Increase of Antibody Response Measured by ELISA 28 Days After the Second Vaccination, 180 Days After the First Vaccination and 28 Days After the Third Vaccination as Compared to Baseline
Description: Geometric mean of fold increase of antibody response measured by IMMUNOZYM ELISA (VIEU/ml) and Enzygnost ELISA (U/ml) from day 0 to specified timeframe. Here, "Number Analyzed" signifies number of participants who were evaluable at the specified timeframe for the specified ELISA assay.
Time Frame: 28 days after Vaccination 2, 180 days after Vaccination 1, 28 days after Vaccination 3
Population: mITT population included eligible participants who fulfilled all inclusion and exclusion criteria, received first and second vaccination, had no positive baseline values in ELISA (IMMUNOZYM FSME ELISA and Enzygnost TBE ELISA) and NT, had immunogenicity measurements available at baseline and 28 days after the second vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 149 | 152
fold rise
  IMMUNOZYM: 180 Days after Vaccination 1: number analyzed (Participants) | 142 | 147
  IMMUNOZYM: 180 Days after Vaccination 1 | 31.6 [26.8 to 37.2] | 9.5 [8.1 to 11]
  IMMUNOZYM: 28 Days after Vaccination 2: number analyzed (Participants) | 143 | 149
  IMMUNOZYM: 28 Days after Vaccination 2 | 193.7 [163 to 230.1] | 39.9 [32.5 to 49]
  IMMUNOZYM: 28 Days after Vaccination 3: number analyzed (Participants) | 141 | 146
  IMMUNOZYM: 28 Days after Vaccination 3 | 719.9 [591.5 to 876.3] | 620.9 [479.7 to 803.6]
  Enzygnost: 180 Days after Vaccination 1: number analyzed (Participants) | 148 | 149
  Enzygnost: 180 Days after Vaccination 1 | 9.5 [8.2 to 11] | 5.3 [4.5 to 6.3]
  Enzygnost: 28 Days after Vaccination 2: number analyzed (Participants) | 149 | 151
  Enzygnost: 28 Days after Vaccination 2 | 32.5 [30.4 to 34.8] | 18.7 [16.3 to 21.5]
  Enzygnost: 28 Days after Vaccination 3: number analyzed (Participants) | 147 | 148
  Enzygnost: 28 Days after Vaccination 3 | 135.8 [115.3 to 160] | 134.6 [106.7 to 169.9]

8. Secondary Outcome: Frequency and Severity of Systemic Reactions Occurring After First Vaccination
Description: Systemic symptoms included headache, nausea, vomiting, muscle pain, joint pain, swelling of the lymph nodes, loss of appetite and changes in sleeping behavior in all age strata; restlessness in children 1 to 2 years of age; malaise and fatigue in participants 3 to 11 years of age as collected in participant diary. Number of participants with systemic reactions according to severity after first vaccination were reported.
Time Frame: Within 28 days after Vaccination 1
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 150 | 152
participants
  Systemic reactions: None | 136 [6.8 to 9.1] | 134 [4.2 to 5.8]
  Systemic reactions: Mild | 13 [39.5 to 55.8] | 15 [19.4 to 28.8]
  Systemic reactions: Moderate | 1 [98.5 to 115.5] | 3 [94.6 to 113.2]
  Systemic reactions: Severe | 0 | 0

9. Secondary Outcome: Frequency and Severity of Systemic Reactions Occurring After Second Vaccination
Description: Systemic symptoms included headache, nausea, vomiting, muscle pain, joint pain, swelling of the lymph nodes, loss of appetite and changes in sleeping behavior in all age strata; restlessness in children 1 to 2 years of age; malaise and fatigue in participants 3 to 11 years of age as collected in participant diary. Number of participants with systemic reactions according to severity after second vaccination were reported.
Time Frame: Within 28 days after Vaccination 2
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 150 | 152
participants
  Systemic reactions: None | 143 [6.8 to 9.1] | 144 [4.2 to 5.8]
  Systemic reactions: Mild | 7 [39.5 to 55.8] | 8 [19.4 to 28.8]
  Systemic reactions: Moderate | 0 [98.5 to 115.5] | 0 [94.6 to 113.2]
  Systemic reactions: Severe | 0 | 0

10. Secondary Outcome: Frequency and Severity of Systemic Reactions Occurring After Third Vaccination
Description: Systemic symptoms included headache, nausea, vomiting, muscle pain, joint pain, swelling of the lymph nodes, loss of appetite and changes in sleeping behavior in all age strata; restlessness in children 1 to 2 years of age; malaise and fatigue in participants 3 to 11 years of age as collected in participant diary. Number of participants with systemic reactions according to severity after third vaccination were reported. Here, "number of participants analyzed" signifies those participants who received FSME-IMMUN or Encepur during the first and second vaccination and received FSME-IMMUN at Day 360 as third vaccination.
Time Frame: Within 28 days after Vaccination 3
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- FSME-IMMUN: It Included participants who received FSME-IMMUN or Encepur during the first and second vaccination and received FSME-IMMUN at Day 360 as third vaccination.
Arm/Group | FSME-IMMUN
Number analyzed (Participants) | 298
participants
  Systemic reactions: None | 282 [6.8 to 9.1]
  Systemic reactions: Mild | 15 [39.5 to 55.8]
  Systemic reactions: Moderate | 1 [98.5 to 115.5]
  Systemic reactions: Severe | 0

11. Secondary Outcome: Frequency and Severity of Injection Site Reactions Occurring After the First Vaccination
Description: Injection site reactions included swelling, induration, redness, injection site pain and tenderness, ecchymosis and hematoma as collected in participant diary. Number of participants with injection site reactions according to severity after first vaccination were reported.
Time Frame: Within 6 days of Vaccination 1
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 150 | 152
participants
  None | 131 [6.8 to 9.1] | 108 [4.2 to 5.8]
  Unknown | 1 [39.5 to 55.8] | 0 [19.4 to 28.8]
  Mild | 18 [98.5 to 115.5] | 41 [94.6 to 113.2]
  Moderate | 0 | 3
  Severe | 0 | 0

12. Secondary Outcome: Frequency and Severity of Injection Site Reactions Occurring After the Second Vaccination
Description: Injection site reactions included swelling, induration, redness, injection site pain and tenderness, ecchymosis and hematoma as collected in participant diary. Number of participants with injection site reactions according to severity after second vaccination were reported.
Time Frame: Within 6 days of Vaccination 2
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 150 | 152
participants
  None | 137 [6.8 to 9.1] | 118 [4.2 to 5.8]
  Mild | 12 [98.5 to 115.5] | 27 [94.6 to 113.2]
  Moderate | 1 | 7
  Severe | 0 | 0

13. Secondary Outcome: Frequency and Severity of Injection Site Reactions Occurring After the Third Vaccination
Description: Injection site reactions included swelling, induration, redness, injection site pain and tenderness, ecchymosis and hematoma as collected in participant diary. Number of participants with injection site reactions according to severity after third vaccination were reported. Here, "number of participants analyzed" signifies those participants who received FSME-IMMUN or Encepur during the first and second vaccination and received FSME-IMMUN at Day 360 as third vaccination.
Time Frame: Within 6 days of Vaccination 3
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | FSME-IMMUN
Number analyzed (Participants) | 298
participants
  None | 249 [6.8 to 9.1]
  Mild | 43 [39.5 to 55.8]
  Moderate | 4 [98.5 to 115.5]
  Severe | 2

14. Secondary Outcome: Frequency and Severity of Adverse Events (AE) Observed Before the Third Vaccination
Description: An AE was any untoward medical occurrence in a participants who received study vaccination without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study vaccine and up to one month after last dose that were absent before treatment or that worsened relative to pre-treatment state. Number of participants with serious and non-serious adverse events according to severity before third vaccination were reported.
Time Frame: Part A: Within 28 days after Vaccination 1 and Vaccination 2, Part B: 28 days after Vaccination 2 to before Vaccination 3
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | FSME-IMMUN | Encepur
Number analyzed (Participants) | 150 | 152
participants
  Non-Serious AE: within 28 days after Vaccination 1 | 57 [6.8 to 9.1] | 80 [4.2 to 5.8]
  Serious AE: within 28 days after Vaccination 1 | 1 [39.5 to 55.8] | 0 [19.4 to 28.8]
  Non-Serious AE: within 28 days after Vaccination 2 | 42 [98.5 to 115.5] | 66 [94.6 to 113.2]
  Serious AE: within 28 days after Vaccination 2 | 0 | 0
  Non-Serious AE:after Part A to before Vaccination3 | 97 | 102
  Serious AE: after Part A to before Vaccination 3 | 6 | 10

15. Secondary Outcome: Frequency and Severity of Adverse Events (AE) Observed After the Third Vaccination
Description: An AE was any untoward medical occurrence in a participants who received study vaccination without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability / incapacity; congenital anomaly. Treatment-emergent are events between first dose of study vaccine and up to one month after last dose that were absent before treatment or that worsened relative to pre-treatment state. Number of participants with serious and non-serious adverse events according to severity after third vaccination were reported. Here, "number of participants analyzed" signifies those participants who received FSME-IMMUN or Encepur during the first and second vaccination and received FSME-IMMUN at Day 360 as third vaccination.
Time Frame: Within 28 days after Vaccination 3
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | FSME-IMMUN
Number analyzed (Participants) | 298
participants
  Non-Serious AE: within 28 days after Vaccination 3 | 102 [6.8 to 9.1]
  Serious AE: within 28 days after Vaccination 3 | 0 [39.5 to 55.8]

ADVERSE EVENTS:
Time Frame: Part A: Within 28 days after Vaccination 1 and Vaccination 2, Part B: 28 days after Vaccination 2 to before the Vaccination 3, within 28 days after Vaccination 3
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included AEs collected in participant diary (local and systemic reactions for FSME-IMMUN) and AEs were documented in participant diary (non-systematic assessment).
Groups:
- Part A (1-2 Years of Age) FSME-IMMUN: After Vaccination 1: Participants aged 1 - 2 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 0, assessed after first vaccination.
- Part A (1-2 Years of Age) FSME-IMMUN: After Vaccination 2: Participants aged 1 - 2 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 28, assessed after second vaccination.
- Part B (1-2 Years of Age) FSME-IMMUN: Before Vaccination 3: Participants aged 1 - 2 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 0 and 28, assessed 28 Days after the second vaccination to prior to third vaccination.
- Part A (3-6 Years of Age) FSME-IMMUN: After Vaccination 1: Participants aged 3 - 6 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 0, assessed after first vaccination.
- Part A (3-6 Years of Age) FSME-IMMUN: After Vaccination 2: Participants aged 3 - 6 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 28, assessed after second vaccination.
- Part B (3-6 Years of Age) FSME-IMMUN: Before Vaccination 3: Participants aged 3 - 6 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 0 and 28, assessed 28 Days after the second vaccination to prior to third vaccination.
- Part A (7-11 Years of Age) FSME-IMMUN: After Vaccination 1: Participants aged 7 - 11 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 0, assessed after first vaccination.
- Part A (7-11 Years of Age) FSME-IMMUN: After Vaccination 2: Participants aged 7 - 11 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 28, assessed after second vaccination.
- Part B (7-11 Years of Age) FSME-IMMUN: Before Vaccination 3: Participants aged 7 - 11 years who received single dose of 0.25 mL FSME-IMMUN Junior (FSME-IMMUN) suspension at Day 0 and 28, assessed 28 Days after the second vaccination to prior to third vaccination.
- Part A (1-2 Years of Age) Encepur: After Vaccination 1: Participants aged 1 - 2 years who received single dose of Encepur Children (Encepur) suspension at Day 0, assessed after first vaccination.
- Part A (1-2 Years of Age) Encepur: After Vaccination 2: Participants aged 1 - 2 years who received single dose of Encepur Children (Encepur) suspension at Day 28, assessed after second vaccination.
- Part B (1-2 Years of Age) Encepur: Before Vaccination 3: Participants aged 1 - 2 years who received single dose of Encepur Children (Encepur) suspension at Day 0 and 28, assessed 28 Days after the second vaccination to prior to third vaccination.
- Part A (3-6 Years of Age) Encepur: After Vaccination 1: Participants aged 3 - 6 years who received single dose of Encepur Children (Encepur) suspension at Day 0, assessed after first vaccination.
- Part A (3-6 Years of Age) Encepur: After Vaccination 2: Participants aged 3 - 6 years who received single dose of Encepur Children (Encepur) suspension at Day 28, assessed after second vaccination.
- Part B (3-6 Years of Age) Encepur: Before Vaccination 3: Participants aged 3 - 6 years who received single dose of Encepur Children (Encepur) suspension at Day 0 and 28, assessed 28 Days after the second vaccination to prior to third vaccination.
- Part A (7-11 Years of Age) Encepur: After Vaccination 1: Participants aged 7 - 11 years who received single dose of Encepur Children (Encepur) suspension at Day 0, assessed after first vaccination.
- Part A (7-11 Years of Age) Encepur: After Vaccination 2: Participants aged 7 - 11 years who received single dose of Encepur Children (Encepur) suspension at Day 28, assessed after second vaccination.
- Part B (7-11 Years of Age) Encepur: Before Vaccination 3: Participants aged 7 - 11 years who received single dose of Encepur Children (Encepur) suspension at Day 0 and 28, assessed 28 Days after the second vaccination to prior to third vaccination.
- Part B (1-2 Years of Age) FSME-IMMUN: After Vaccination 3: Participants aged 1 - 2 years who received either FSME-IMMUN or Encepur during the first and second vaccination, received FSME-IMMUN Junior (FSME-IMMUN) at Day 360 as third vaccination. Assessment of AEs was done after the third vaccination.
- Part B (3-6 Years of Age) FSME-IMMUN: After Vaccination 3: Participants aged 3 - 6 years who received either FSME-IMMUN or Encepur during the first and second vaccination, received FSME-IMMUN Junior (FSME-IMMUN) at Day 360 as third vaccination. Assessment of AEs was done after the third vaccination.
- Part B (7-11 Years of Age) FSME-IMMUN: After Vaccination 3: Participants aged 7 - 11 years who received either FSME-IMMUN or Encepur during the first and second vaccination, received FSME-IMMUN Junior (FSME-IMMUN) at Day 360 as third vaccination. Assessment of AEs was done after the third vaccination.
Arm/Group | Part A (1-2 Years of Age) FSME-IMMUN: After Vaccination 1 | Part A (1-2 Years of Age) FSME-IMMUN: After Vaccination 2 | Part B (1-2 Years of Age) FSME-IMMUN: Before Vaccination 3 | Part A (3-6 Years of Age) FSME-IMMUN: After Vaccination 1 | Part A (3-6 Years of Age) FSME-IMMUN: After Vaccination 2 | Part B (3-6 Years of Age) FSME-IMMUN: Before Vaccination 3 | Part A (7-11 Years of Age) FSME-IMMUN: After Vaccination 1 | Part A (7-11 Years of Age) FSME-IMMUN: After Vaccination 2 | Part B (7-11 Years of Age) FSME-IMMUN: Before Vaccination 3 | Part A (1-2 Years of Age) Encepur: After Vaccination 1 | Part A (1-2 Years of Age) Encepur: After Vaccination 2 | Part B (1-2 Years of Age) Encepur: Before Vaccination 3 | Part A (3-6 Years of Age) Encepur: After Vaccination 1 | Part A (3-6 Years of Age) Encepur: After Vaccination 2 | Part B (3-6 Years of Age) Encepur: Before Vaccination 3 | Part A (7-11 Years of Age) Encepur: After Vaccination 1 | Part A (7-11 Years of Age) Encepur: After Vaccination 2 | Part B (7-11 Years of Age) Encepur: Before Vaccination 3 | Part B (1-2 Years of Age) FSME-IMMUN: After Vaccination 3 | Part B (3-6 Years of Age) FSME-IMMUN: After Vaccination 3 | Part B (7-11 Years of Age) FSME-IMMUN: After Vaccination 3
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50 | 1/50 | 0/51 | 0/51 | 3/51 | 0/49 | 0/49 | 2/48 | 0/50 | 0/50 | 4/50 | 0/51 | 0/51 | 3/51 | 0/51 | 0/51 | 3/51 | 0/99 | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 17/50 | 13/50 | 37/50 | 15/51 | 11/51 | 30/51 | 14/49 | 10/49 | 30/48 | 25/50 | 13/50 | 39/50 | 33/51 | 19/51 | 33/51 | 30/51 | 26/51 | 30/51 | 23/99 | 29/100 | 30/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (1-2 Years of Age) FSME-IMMUN: After Vaccination 1 (N=50) | Part A (1-2 Years of Age) FSME-IMMUN: After Vaccination 2 (N=50) | Part B (1-2 Years of Age) FSME-IMMUN: Before Vaccination 3 (N=50) | Part A (3-6 Years of Age) FSME-IMMUN: After Vaccination 1 (N=51) | Part A (3-6 Years of Age) FSME-IMMUN: After Vaccination 2 (N=51) | Part B (3-6 Years of Age) FSME-IMMUN: Before Vaccination 3 (N=51) | Part A (7-11 Years of Age) FSME-IMMUN: After Vaccination 1 (N=49) | Part A (7-11 Years of Age) FSME-IMMUN: After Vaccination 2 (N=49) | Part B (7-11 Years of Age) FSME-IMMUN: Before Vaccination 3 (N=48) | Part A (1-2 Years of Age) Encepur: After Vaccination 1 (N=50) | Part A (1-2 Years of Age) Encepur: After Vaccination 2 (N=50) | Part B (1-2 Years of Age) Encepur: Before Vaccination 3 (N=50) | Part A (3-6 Years of Age) Encepur: After Vaccination 1 (N=51) | Part A (3-6 Years of Age) Encepur: After Vaccination 2 (N=51) | Part B (3-6 Years of Age) Encepur: Before Vaccination 3 (N=51) | Part A (7-11 Years of Age) Encepur: After Vaccination 1 (N=51) | Part A (7-11 Years of Age) Encepur: After Vaccination 2 (N=51) | Part B (7-11 Years of Age) Encepur: Before Vaccination 3 (N=51) | Part B (1-2 Years of Age) FSME-IMMUN: After Vaccination 3 (N=99) | Part B (3-6 Years of Age) FSME-IMMUN: After Vaccination 3 (N=100) | Part B (7-11 Years of Age) FSME-IMMUN: After Vaccination 3 (N=99)
HYPOSPADIAS (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CRYPTORCHISM (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EUSTACHIAN TUBE DISORDER (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HERPANGINA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACUTE TONSILLITIS (Infections and infestations) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FOREIGN BODY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACQUIRED PHIMOSIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ADENOIDAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ORCHIDOPEXY (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (1-2 Years of Age) FSME-IMMUN: After Vaccination 1 (N=50) | Part A (1-2 Years of Age) FSME-IMMUN: After Vaccination 2 (N=50) | Part B (1-2 Years of Age) FSME-IMMUN: Before Vaccination 3 (N=50) | Part A (3-6 Years of Age) FSME-IMMUN: After Vaccination 1 (N=51) | Part A (3-6 Years of Age) FSME-IMMUN: After Vaccination 2 (N=51) | Part B (3-6 Years of Age) FSME-IMMUN: Before Vaccination 3 (N=51) | Part A (7-11 Years of Age) FSME-IMMUN: After Vaccination 1 (N=49) | Part A (7-11 Years of Age) FSME-IMMUN: After Vaccination 2 (N=49) | Part B (7-11 Years of Age) FSME-IMMUN: Before Vaccination 3 (N=48) | Part A (1-2 Years of Age) Encepur: After Vaccination 1 (N=50) | Part A (1-2 Years of Age) Encepur: After Vaccination 2 (N=50) | Part B (1-2 Years of Age) Encepur: Before Vaccination 3 (N=50) | Part A (3-6 Years of Age) Encepur: After Vaccination 1 (N=51) | Part A (3-6 Years of Age) Encepur: After Vaccination 2 (N=51) | Part B (3-6 Years of Age) Encepur: Before Vaccination 3 (N=51) | Part A (7-11 Years of Age) Encepur: After Vaccination 1 (N=51) | Part A (7-11 Years of Age) Encepur: After Vaccination 2 (N=51) | Part B (7-11 Years of Age) Encepur: Before Vaccination 3 (N=51) | Part B (1-2 Years of Age) FSME-IMMUN: After Vaccination 3 (N=99) | Part B (3-6 Years of Age) FSME-IMMUN: After Vaccination 3 (N=100) | Part B (7-11 Years of Age) FSME-IMMUN: After Vaccination 3 (N=99)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CRYPTORCHISM (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MIDDLE EAR INFLAMMATION (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
THYROIDITIS (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
FATIGUE (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 3
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 3 | 2 | 0 | 3 | 4 | 0 | 1 | 4 | 4
INJECTION SITE HAEMATOMA (General disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 3
INJECTION SITE HAEMORRHAGE (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
INJECTION SITE INDURATION (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 3 | 3 | 0 | 4 | 2 | 0 | 0 | 3 | 6
INJECTION SITE PAIN (General disorders) | 1 | 2 | 0 | 3 | 3 | 0 | 10 | 5 | 0 | 4 | 1 | 0 | 10 | 6 | 0 | 24 | 24 | 0 | 2 | 13 | 27
INJECTION SITE PRURITUS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
INJECTION SITE SWELLING (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 7
MALAISE (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 9 | 2 | 0 | 4 | 3 | 3 | 4 | 1 | 5 | 9 | 3 | 0 | 5 | 3 | 2 | 4 | 2 | 3 | 3 | 8 | 0
TENDERNESS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ALLERGIC OEDEMA (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MULTIPLE ALLERGIES (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ACUTE TONSILLITIS (Infections and infestations) | 0 | 0 | 5 | 1 | 0 | 4 | 0 | 0 | 1 | 2 | 1 | 5 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 0
BACTERIAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 3 | 2 | 1 | 0 | 0 | 2 | 4 | 1 | 0 | 4 | 0 | 2 | 0
BRONCHITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVITIS INFECTIVE (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
EAR INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ENTEROBIASIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
ERYTHEMA INFECTIOSUM (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
EXANTHEMA SUBITUM (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 3 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
GENITAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HERPANGINA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
IMPETIGO (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
LARYNGITIS (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 2 | 2 | 1 | 7 | 0 | 1 | 6 | 0 | 0 | 5 | 1 | 1 | 7 | 3 | 1 | 7 | 0 | 2 | 3
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 1 | 3 | 8 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 8 | 1 | 1 | 2 | 0 | 0 | 0 | 5 | 2 | 0
OTITIS MEDIA ACUTE (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PARONYCHIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PAROTITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 9 | 1 | 0 | 0 | 0 | 1 | 5 | 1 | 0 | 5 | 0 | 6 | 1
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PSEUDOCROUP (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
SCARLET FEVER (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
TONSILLITIS (Infections and infestations) | 0 | 2 | 10 | 0 | 0 | 2 | 1 | 0 | 5 | 3 | 0 | 12 | 0 | 0 | 3 | 1 | 1 | 2 | 3 | 2 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TRACHEITIS (Infections and infestations) | 1 | 2 | 17 | 0 | 0 | 7 | 0 | 0 | 1 | 1 | 3 | 13 | 0 | 2 | 6 | 0 | 0 | 0 | 5 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
VARICELLA (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 5 | 0 | 0 | 0 | 3 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 4 | 2 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 3 | 2 | 0 | 0
VIRAL RASH (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VIRAL TONSILLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEAT STROKE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MOUTH INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OPEN WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BODY TEMPERATURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEART RATE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OBESITY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
UNDERWEIGHT (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 3 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 5 | 2 | 1 | 0 | 3 | 7
ATTENTION DEFICIT/HYPERACTIVITY DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RESTLESSNESS (Psychiatric disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SLEEP DISORDER (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
TIC (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MICTURITION DISORDER (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ACQUIRED PHIMOSIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BALANITIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ADENOIDAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 2 | 0 | 1 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TRACHEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TOOTH EXTRACTION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.